CLINICAL TRIAL: NCT00728962
Title: A Prospective, Observational Study of Osseotite Certain IOL (Immediate Occlusal Loading) Implants in Immediate Occlusal Loading of Short Span Fixed Restorations
Brief Title: A Study of Osseotite Certain Prevail Implants Used to Support Short Fixed Bridges With Immediate Occlusal Loading.
Acronym: Fireball
Status: Completed | Type: Observational
Sponsor: ZimVie (Industry)
Responsible Party: Sponsor
Other Study IDs: 2208
Record Dates: First submitted 2008-08-01; First posted 2008-08-06 (Estimated); Results first posted 2010-02-05 (Estimated); Last update posted 2022-04-19 (Actual); Status verified 2022-03

CONDITIONS: Partial Edentulism; Tooth Disease
Keywords: dental implants; Osseotite Certain Prevail; multicenter; observational; clinical study; partial edentulism; single stage; immediate occlusal loading; crestal bone level; short fixed bridge
MeSH Terms: conditions — Tooth Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This prospective, multicenter study evaluates the performance of the Osseotite Prevail implant when to support a short fixed bridge with immediate occlusal loading, providing the patient with the use of a temporary prosthesis until the final prosthesis is made.

Study (null) hypothesis: This is an observational study in which no concurrent control group will be observed. Results of the study will be compared with the performance of other Osseotite implants from published Osseotite multicenter studies.

DETAILED DESCRIPTION:
This is a prospective, observational study in which all the patients will have implants placed and a provisional prosthesis attached within 24 hours of implant surgery. Each restorative case will consist of a posterior short span fixed bridge of four implants or less. The final prosthesis will be placed within five months or implant placement surgery. Overall success will be determined on the basis of procedural success, prosthesis success, and implant success.

ELIGIBILITY:
Inclusion Criteria:

* patients of either sex and of any race, 18 years of age or older
* patients for whom the decision has already been made to use dental implants for treating partial edentulism in the posterior mandible or maxilla using a short span fixed prosthesis of two to four units
* patients must be physically able to tolerate conventional surgical and restorative procedures
* requirements for implant placement include: at least 1mm bone will be available at the buccal and lingual aspect of the implant and at least 1mm of bone below the apex
* patients must agree to return to the clinic for each study follow-up visit
* requirements for prosthetic fabrication include: bone width at least 6mm and a bone height of at least 11mm

Exclusion Criteria:

* patients with active infection or severe inflammation in the areas intended for implant placement
* patients with a >10 cigarettes / day smoking habit
* patients with uncontrolled diabetes or metabolic bone disease
* patients with a history of therapeutic radiation to the head
* patients in need of bone grafting at the site of the intended study implant; if at the time of surgery some lateral voids need to be filled this is acceptable and does not exclude the patient from the analysis
* patients who are known to be pregnant
* patients with para-functional habits with evidence of severe bruxing or clenching
* placement of implants into sites with less than sixteen weeks of post-extraction healing; for 3-4 unit cases one implant site may have less than sixteen weeks of healing prior to implant placement
* type III or IV bone characteristics of the intended implant sites
* inter-arch distance of less than 7mm (planned location of implant seating platform to the apposing occlusal landmark)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: These will be patients who are otherwise seeking dental implant therapy and belong to the study centers' standard patient population.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2005-03; Primary Completion 2006-05 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hessam Nowzari, DDS, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Each site endeavored to enroll a maximum of 15 patients, with enrollment efforts beginning in March 2005. Enrollment period remained open at all sites until April 2006. Three participating sites are Universities and four are private practices.
Pre-assignment Details: Pre-treatment included a screening visit(enroll those meeting all study inclusion criteria), signing informed consent, and pre-surgical data collection. Within 48hrs., impressions of the patient's treatment areas are taken for making a temporary prosthesis. Patients are then scheduled for implant placement surgery.
Groups:
- Osseotite Certain Prevail Implant: Internal connection implant with an expanded platform and lateralization with a tapered apex
Period: Implant Placement Surgery
Arm/Group | Osseotite Certain Prevail Implant
Started | 75
Completed | 65
Not Completed | 10
Not completed — Adverse Event | 8
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 1
Period: Permanent Prosthesis Placement
Arm/Group | Osseotite Certain Prevail Implant
Started | 65
Completed | 62
Not Completed | 3
Not completed — Adverse Event | 3
Period: One Year Post Placement Follow-up
Arm/Group | Osseotite Certain Prevail Implant
Started | 62
Completed | 62
Not Completed | 0
Period: Two Year Post Placement Follow-up
Arm/Group | Osseotite Certain Prevail Implant
Started | 62
Completed | 59
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Osseotite Certain Prevail Implant
Number analyzed (Participants) | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 62
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 39
Region of Enrollment [Number; unit: participants]
  United States | 22
  Italy | 17
  Netherlands | 7
  France | 16
  Germany | 13

OUTCOME MEASURES:

1. Primary Outcome: Patients With Implants Achieving Osseous Integration
Description: Patients receiving test implant(s) will achieve integration success (implant show no signs of mobility) of the implant at the time of analysis.
Time Frame: 1 year
Population: total number of patients enrolled in the study was used for primary outcome analysis
Measure: Number; unit: participants
Arm/Group | Osseotite Certain Prevail Implant
Number analyzed (Participants) | 75
participants | 59

2. Secondary Outcome: Crestal Bone Regression
Time Frame: four years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event reports are collected from day 1 to present; 4 years of study duration to date.
Description: Adverse event data is collected during each study event visit the patient is seen for.
Arm/Group | Osseotite Certain Prevail Implant
Serious Adverse Events (participants affected / at risk) | 0/75
Other Adverse Events (participants affected / at risk) | 11/75
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Osseotite Certain Prevail Implant (N=75)
Loss of integration of implant (Surgical and medical procedures) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall furnish SPONSOR with a copy of any proposed publication thirty (30) days prior to submission for publication for review and comment. SPONSOR may request PI to delay publishing such proposed publication for a maximum of an additional sixty (60) days in order to protect the potential patentability of any invention described therein.